CLINICAL TRIAL: NCT01507610
Title: An Open-Label, Single-Dose, Randomized, Crossover Study to Compare the Bioavailability of the Intranasal Administration of 20 mg OPTINOSE SUMATRIPTAN With 20 mg IMITREX® (Sumatriptan) Nasal Spray, 100 mg IMITREX® (Sumatriptan) Oral Tablet and 6 mg IMITREX® (Sumatriptan) Subcutaneous Injection in Healthy Subjects
Brief Title: Bioavailability Study to Compare OPTINOSE SUMATRIPTAN With IMITREX® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OPN-SUM-1302
Record Dates: First submitted 2012-01-04; First posted 2012-01-11 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-01

CONDITIONS: Migraine
Keywords: sumatriptan; bioavailability
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Investigational (Experimental): OPTINOSE SUMATRIPTAN, single dose of 20 mg intranasally (10 mg to each nostril).
  Interventions: Drug: Sumatriptan
- IMITREX Nasal Spray (Active Comparator): IMITREX® (sumatriptan) Nasal Spray, single dose of 20 mg intranasally (20 mg to one nostril).
  Interventions: Drug: Sumatriptan
- IMITREX Oral Tablet (Active Comparator): IMITREX® (sumatriptan) Oral Tablet, single dose of 100 mg, administered orally with 240 mL water.
  Interventions: Drug: Sumatriptan
- IMITREX Subcutaneous Injection (Active Comparator): IMITREX® (sumatriptan) Subcutaneous Injection, single dose of 6 mg injected subcutaneously in the abdomen.
  Interventions: Drug: Sumatriptan

INTERVENTIONS:
Drug: Sumatriptan — To compare the single-dose pharmacokinetics (PK) and relative bioavailability of intranasal administration of 20 mg OPTINOSE SUMATRIPTAN with 20 mg IMITREX® (sumatriptan) Nasal Spray, 100 mg IMITREX® (sumatriptan) Oral Tablet, and 6 mg IMITREX® (sumatriptan) Subcutaneous Injection, in healthy subjects.

SUMMARY:
The purpose of this study is:

* To compare the single-dose pharmacokinetics (PK) of intranasal administration of 20 mg OPTINOSE SUMATRIPTAN with 20 mg IMITREX® (sumatriptan) Nasal Spray, 100 mg IMITREX® (sumatriptan) Oral Tablet, and 6 mg IMITREX® (sumatriptan) Subcutaneous Injection, in healthy subjects.
* To estimate the relative bioavailability of single-dose intranasal administration of 20 mg OPTINOSE SUMATRIPTAN, 20 mg IMITREX® (sumatriptan) Nasal Spray, and 100 mg IMITREX® (sumatriptan) Oral Tablet compared to a single-dose of 6 mg IMITREX® (sumatriptan) Subcutaneous Injection, in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ages 18 to 55 years, inclusive, at screening.
* Healthy with no clinically relevant abnormalities in the opinion of the Investigator as determined by medical history, physical examination, blood chemistry, hematology, including complete blood count, urinalysis, vital signs, and ECG.
* Have a BMI of 18-32 kg/m2, inclusive, and a body weight of not less than 50 kg.
* For females of childbearing potential: either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using one of the following acceptable birth control methods:

  * intrauterine device in place for at least 3 months prior to the first dose and throughout the study.
  * barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study.
  * surgical sterilization of the partner (vasectomy for 6 months minimum).
  * hormonal contraceptives for at least 3 months prior to the first dose of the study and throughout the study.
  * Female subjects who claim to be sexually inactive, but become sexually active during the course of the study must agree to use a barrier method (e.g. condom, diaphragm) with spermicide from the time of the start of sexual activity through completion of the study.
  * In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for the whole duration of the study.
* Females of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to Day 1:

  * bilateral tubal ligation
  * hysterectomy
  * bilateral oophorectomy or be postmenopausal with amenorrhea for at least 1 year prior to Day 1 and follicle stimulating hormone (FSH) serum levels ≥ 40 mIU/mL.
* Women of child-bearing potential must have a negative serum beta-human chorionic gonadotropin at the screening visit and at each check-in prior to dosing.
* Agree to abstain from alcohol intake 48 hours before each administration of study agent and during inpatient portion of the study.
* Agree to limit caffeine/methylxanthine (eg, coffee, tea, chocolate, or caffeine-containing soft drinks) intake to less than 300 mg/day for 7 days prior to and for the duration of the study (300 mg of caffeine is equal to approximately 3 cups of coffee or 6 cola drinks), with no intake from 24 hours before dosing and throughout confinement.
* Agree not to consume food or beverages containing, grapefruit or grapefruit juice, Seville oranges, or quinine (e.g. tonic water) 72 hours prior to study Day -1 until after the last PK sample is collected.
* Agree not to consume food containing poppy seeds during the study.
* Have verified airflow through both nostrils and an ability to close the soft palate.
* Must be able to use the OptiNose device correctly.
* Subjects must understand English and have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Be willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Currently have or have a history of disease or dysfunction of the pulmonary, cardiovascular, endocrine, hematologic, neurological, immune, gastrointestinal, genitourinary, or other body system that is clinically significant in the opinion of the Investigator.
* Have evidence of any chronic medical conditions requiring prescription medications (eg, hypertension or diabetes).
* Have a history of migraines.
* History of hypersensitivity or allergies to any drug compound, including sumatriptan, any of its components or sulphonamides.
* Have had a major or traumatic surgery within 12 weeks prior to screening, pre-planned surgery or procedures that would interfere with the conduct of the study.
* Have an acute illness within 7 days prior to study agent administration or have had a major illness or hospitalization within 1 month prior to study agent administration.
* Have clinically significant findings on screening ECG.
* Have a recent history (within 1 previous year) of alcohol or drug abuse.
* History of smoking or use of nicotine-containing substances within the previous 2 months.
* Have abnormal values for hematology, clinical chemistry, or urinalysis at screening or check-in considered clinically significant by the Investigator.
* Have a positive serology test for HIV antibodies, HBsAg, or hepatitis C virus antibody (anti-HCV) at screening.
* Have a positive urine drug screen for ethanol or substances of abuse including cocaine, cannabinoids, phencyclidine, amphetamines, benzodiazepines, barbiturates, opiates, propoxyphene, and methadone at screening and each check-in.
* Have a haemoglobin level below the lower limit of normal at screening.
* Have donated blood or experienced significant blood loss (volume > 500 mL) within 3 months prior to screening, or is planning to donate within 2 months after completion of the study.
* Use of drug metabolizing enzyme (CYP-450) inducers within 28 days prior to dosing or inhibitors within 14 days prior to dosing (refer to Appendix 1).
* Use of any monoamine oxidase inhibitors (MAOI) within 28 days prior to dosing.
* Use of any prescription medications/products, except hormonal contraceptives, within 14 days prior to study entry.
* Use of any OTC, nonprescription preparation (including minerals and phytotherapeutic/herbal/plant-derived preparations), within 14 days prior to study entry, with the exception of ibuprofen, and acetaminophen used at recommended doses. For acetaminophen, a maximum of 1500 mg per day and no more than 3 g per week, will be allowed for the treatment of headache or other pain.
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 4 weeks prior to dosing, or plan to participate in an investigational drug study less than 1 month after completion of the study.
* A recent febrile illness within 3 days of the start of the study drug intake on Day 1.
* If a woman, must not be breast-feeding or planning to become pregnant during the study.
* Must refrain from physical activity (jogging, strenuous exercise of all types), and sunbathing while confined to the study center and 48 hours before admission to the study center.
* Reports or exhibits abnormalities regarding the sense of smell and/or taste.
* Reports a temporary loss of or abnormality of sense of smell and/or taste due to recent (within the 2 weeks prior to Day 1) cold or viral infections.
* Presence of respiratory diseases or known nasal obstruction including allergic rhinitis, nasal septum deviation, polyposis, severe mucosal swelling, nasal ulcers, nasal trauma,or any other reason.
* Have a history of chronic nose bleeds.
* Current nasopharyngeal illness.
* Known velum insufficiency, ie, those with cleft palate and/or structural abnormalities in the soft palate and nasopharynx.
* Any condition that in the opinion of the Investigator would complicate or compromise the study, or the well-being of the subject.
* Is an employee of the Investigator/study center or the Sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameters of sumatriptan following the administration of OPTINOSE SUMATRIPTAN and IMITREX® (sumatriptan). | Measurement of pharmacokinetic parameters of sumatriptan at pre-treatment and at: 2, 5, 10, 15, 20, 25, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hours post treatments.
  The pharmacokinetic parameters AUC0-∞ and Cmax of sumatriptan following the administration of 20 mg OPTINOSE SUMATRIPTAN, 20 mg IMITREX® (sumatriptan) Nasal Spray, 100 mg IMITREX® (sumatriptan) Oral Tablet, and 6 mg IMITREX® (sumatriptan) Subcutaneous Injection.
  • The relative bioavailability (Frel) of sumatriptan following the nasal administration of 20 mg OPTINOSE SUMATRIPTAN, 20 mg IMITREX® (sumatriptan) Nasal Spray, and 100 mg IMITREX® (sumatriptan) Oral Tablet compared to 6 mg IMITREX® (sumatriptan) Subcutaneous Injection.
Bioavailability of sumatriptan following the administration of OPTINOSE SUMATRIPTAN and IMITREX® (sumatriptan). | Measurement of plasma sumatriptan concentrations at pre-treatment and at: 2, 5, 10, 15, 20, 25, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hours post treatments.
  The relative bioavailability (Frel) of sumatriptan following the nasal administration of 20 mg OPTINOSE SUMATRIPTAN, 20 mg IMITREX® (sumatriptan) Nasal Spray, and 100 mg IMITREX® (sumatriptan) Oral Tablet compared to 6 mg IMITREX® (sumatriptan) Subcutaneous Injection.

SECONDARY OUTCOMES:
Sensory attributes of the intranasal OPTINOSE SUMATRIPTAN product and IMITREX® (sumatriptan). | Sensory attributes will be evaluated within 2 minutes after drug administration. The evaluation will be repeated within 5 to 10 minutes after drug administration.
  Sensory attributes of the intranasal OPTINOSE SUMATRIPTAN product, IMITREX® (sumatriptan) Nasal Spray and 100 mg IMITREX® (sumatriptan) Oral Tablet will be evaluated using a 14-item or 4 item Sensory Nasal Spray Evaluation Questionnaire.
Safety Evaluations of the intranasal OPTINOSE SUMATRIPTAN product and IMITREX® | Safety evaluations will be perfromed on days 1, 8, 15, 22, 25 and 32
  Safety evaluation will be based on physical examinations, vital signs, 12-lead electrocardiograms (ECGs), clinical laboratory tests (hematology, serum chemistry and urinalysis), and adverse events (AEs).

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Neptune City, New Jersey, United States

REFERENCES:
- [Derived] Obaidi M, Offman E, Messina J, Carothers J, Djupesland PG, Mahmoud RA. Improved pharmacokinetics of sumatriptan with Breath Powered nasal delivery of sumatriptan powder. Headache. 2013 Sep;53(8):1323-33. doi: 10.1111/head.12167. Epub 2013 Aug 28. PMID 23992438